CLINICAL TRIAL: NCT07388927
Title: Effectiveness of Hirudoid on Ecchymosis After Periorbital Rejuvenation With Botulinum Toxin Type A - A Real-World Multicenter, Prospective, Interventional Study
Brief Title: A Real-World Study on Effect of Hirudoid on Ecchymosis After Treatment of Crow's Feet With Botulinum Toxin Type A
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: DKSH Management (Thailand) Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DKS-HIRUDOID-RWE
Record Dates: First submitted 2025-12-30; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Ecchymosis After Periorbital Rejuvenation With Botulinum Toxin Type A; Crow's Feet Lines; Lateral Canthal Lines, LCL
Keywords: Hirudoid; Botox; botulinum toxin type A injection; Bruising; Periorbital rejuvenation; Ecchymosis; Lateral canthal lines; Crow's feet
MeSH Terms: conditions — Contusions; Ecchymosis | interventions — Hirudoid; Heparinoids; Ointments

STUDY DESIGN:
Intervention Model Description: This will be an intra-individual comparison study, where the study drug will be applied to one side of the face of participants, and the other half of the face will receive no treatment.
  A computer-generated random sheet will be used to assign the right/left side of the face for treatment, to avoid allocation bias and to improve scientific validity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hirudoid (Experimental): All enrolled and eligible participants who are planning to receive botulinum toxin type A for lateral canthal lines will receive the study drug (Hirudoid).
  Interventions: Drug: Hirudoid (heparinoids) ointment, 3mg/g

INTERVENTIONS:
Drug: Hirudoid (heparinoids) ointment, 3mg/g — This study is to observe the effectiveness of Hirudoid on ecchymosis after treatment of Crow's feet with botulinum toxin type A. Hirudoid is a topical treatment that is indicated for the soothing relief of superficial bruising and haematoma. It may potentially reduce the severity (intensity and extent) of bruising, and/or increase the speed of resolution of bruising after periorbital botulinum toxin A injection.
  Hirudoid will be applied to one side of the face (randomized allocation of left or right) for all eligible participants, 30 minutes before the botulinum toxin type A injection procedure, and three times a day, starting 24 hours after the procedure, until post-procedure Day 10.
  A 2 centimetre ribbon of Hirudoid will be applied to the affected area (i.e. the lateral canthal lines injection site), and massaged into skin until absorbed.

SUMMARY:
Botulinum toxin type A (commonly referred to as 'Botox') injections are a treatment that dermatologists regularly use to smoothen wrinkles such as 'Crow's feet', to rejuvenate the skin surrounding the eye (the 'periorbital region'). However, botulinum toxin type A can be associated with injection-site bruising that may take up to 2 weeks to heal.

Hirudoid, an ointment that is applied to the skin, has been shown to reduce the severity of swelling and bruising after facial cosmetic procedures. The objective of this study is to study the effectiveness of Hirudoid in reducing the severity of bruising following the use of botulinum toxin type A for periorbital rejuvenation of Crow's feet in adult patients.

The knowledge gained from this study can help to develop an effective medicated skincare regimen that helps to minimize the complications of botulinum toxin type A and speed up recovery time, which may be of benefit to patients who receive botulinum toxin type A injections for treatment of Crow's feet.

DETAILED DESCRIPTION:
This is an investigator-initiated, real-world, multicenter, prospective, interventional study to assess the effectiveness of topical Hirudoid for both preventing, and reducing the severity (intensity and extent) of ecchymosis after periorbital rejuvenation with botulinum toxin type A. This will be an intra-individual comparison study, where the study drug will be applied to one side of the face, and the other half of the face will receive no treatment.

Planned follow up is up to 10 days with assessments scheduled at Days 1, 2, 5, 7, and 10 post-botulinum toxin type A injection. The total number of mandatory in-person visits would be 2, including a visit on the day of botulinum toxin type A injection (Day 0), and a follow-up visit on Day 7 post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years) undergoing periorbital rejuvenation procedures with botulinum toxin type A (e.g., improvement in the appearance of moderate-to-severe lateral canthal lines)
* Patients willing to participate in the study and return for the scheduled follow-up visit, be photographed as a part of the study procedures, and sign the informed consent form

Exclusion Criteria:

* Known allergy to Hirudoid or any components of Hirudoid
* Known allergy to Botulinum toxin type A
* Previous cosmetic surgery or visible scars in the treatment area
* Severe atrophy or weakness in the target muscles
* Use of local anesthetic prior to Botulinum toxin type A administration
* Current or recent use of anticoagulant or corticosteroid therapy
* Current cigarette smoker
* History of clotting or coagulation disorders
* History of cardiovascular, metabolic, endocrine, liver or renal diseases or any underlying medical condition that may interfere with the study procedures or assessments
* Patients suffering from any psychiatric condition
* Patients taking any agent (e.g., aminoglycoside antibiotics) or suffering from any disorder (e.g., myasthenia gravis, Eaton-Lambert syndrome) that may interfere with neuromuscular function
* Pregnant or lactating women
* Patients unwilling to be photographed or sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Area (extent) of ecchymosis around the eye | Day 7 post-procedure with botulinum toxin type A
  Area (extent) of ecchymosis around the eye with Hirudoid versus 'no treatment' on day 7 post-procedure with botulinum toxin type A for the treatment of lateral canthal lines.
  Patients will be instructed to take daily photographs of both sides of face, which will be shared with clinician and analysed with online software to measure area of bruising using a freehand selection tool to trace the border. Results are to be inputted into the electronic case record form in cm2. A separate independent assessment will take place for each image, by a second physician who is blinded to initial results.

SECONDARY OUTCOMES:
Area (extent) of ecchymosis around the eye | Days 1, 2, 5 and 10 post-procedure with botulinum toxin type A
  Area (extent) of ecchymosis around the eye with Hirudoid versus 'no treatment' on days 1, 2, 5 and 10 post-procedure with botulinum toxin type A, using the methodology described for primary endpoint.
  Patients will be instructed to take daily photographs of both sides of face, which will be shared with clinician and analysed with online software to measure area of bruising using a freehand selection tool to trace the border. Results are to be inputted into the electronic case record form in cm2. A separate independent assessment will take place for each image, by a second physician who is blinded to initial results.
Intensity of ecchymosis around the eye | Days 1, 2, 5, 7 and 10 post-procedure with botulinum toxin type A
  Intensity of ecchymosis around the eye with Hirudoid versus 'no treatment' on days 1, 2, 5, 7 and 10 post-procedure with botulinum toxin type A for the treatment of lateral canthal lines.
  Patients will be instructed to take daily photographs of both sides of face, which will be shared with clinician and analysed against a 5-item scoring system (adapted from Rostami et al. 2020) for assessing the intensity of ecchymosis around the eye, where higher scores indicate greater post-procedure bruising. Rating: 0 (no colour change); 1 (yellowish colour change); 2 (light purple); 3 (dark purple); 4 (very dark purple).
  A separate independent assessment will take place for each image, by a second physician who is blinded to initial results.
Duration (days until resolution) of ecchymosis | Day 1 to Day 10 post-procedure with botulinum toxin type A
  Duration (days until resolution) of ecchymosis with study treatment versus 'no treatment' assessed based on visual assessment by the physician using the using the scoring system adapted from Rostami et al. 2020.
  Patients will be instructed to take daily photographs of both sides of face, which will be shared with clinician and analysed against a 5-item scoring system for assessing the intensity of ecchymosis around the eye, where gradual reduction of ratings indicate resolution. Rating: 0 (no colour change); 1 (yellowish colour change); 2 (light purple); 3 (dark purple); 4 (very dark purple). A separate independent assessment will take place for each image, by a second physician who is blinded to initial results.
Global patient satisfaction | Day 7 post-procedure with botulinum toxin type A
  Global patient satisfaction relating to the impact and outcomes of Hirudoid treatment, evaluated by a 5-point Likert-scale questionnaire (1=very dissatisfied to 5=very satisfied) on day 7 post-procedure.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Day 1 to Day 10 post-procedure with botulinum toxin type A
  Incidence and type of local adverse events will be summarized descriptively using count and percentages for both the arms.

IPD SHARING:
Plan to Share IPD: Yes
Complete data will not be shared with any other institution or personnel in a way which can expose the identity of participating patients. All records identifying the patient will be kept confidential and, to the extent permitted by the applicable laws and/or regulations, will not be made publicly available.
  A summary of the pooled participant study data based on the approved statistical analysis plan, will be shared in the form of an abbreviated clinical study report.
Supporting Information: CSR
Time Frame: Tentative dates available: May 2026 to May 2026 No end date.
Access Criteria: A summary of the pooled participant study data based on the approved statistical analysis plan, will be shared in the form of an abbreviated clinical study report. This clinical study report document will be available to researchers on email request to the corresponding author of the manuscript.